CLINICAL TRIAL: NCT04049578
Title: A Phase Ib, Multicenter, Open-Label, 6-Week Study With a 48-Week Extension to Investigate the Pharmacokinetics, Safety, and Tolerability of Balovaptan in Children Ages 2-4 Years With Autism Spectrum Disorder
Brief Title: A Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Balovaptan in Children With Autism Spectrum Disorder
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recent analysis of Phase II balovaptan data in paediatric ASD did not support the continuation of this study. No new safety concerns were identified.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WP40877
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — balovaptan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Balovaptan (Experimental)
  Interventions: Drug: Balovaptan

INTERVENTIONS:
Drug: Balovaptan — Participants were to receive an oral dose of balovaptan once a day (QD) for a 6-week treatment period, followed by an optional extension period of 48 weeks.

SUMMARY:
This was a Phase Ib, multicenter, open-label study in children 2-4 years old with autism spectrum disorder (ASD) to investigate the pharmacokinetics, safety, and tolerability of an oral dose of balovaptan once a day (QD). The study was to consists of a 6-week treatment period to evaluate the pharmacokinetics of balovaptan in 2 to 4 year old children followed by an optional extension period of 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ASD according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for ASD. Diagnostics will be performed by a team of autism experts and confirmed by Autism Diagnostic Observation ScheduleTM, Second Edition (ADOS-2) criteria. The DSM-5 criteria for diagnosis of autism must be met with the highest confidence in the opinion of the investigator. Children with ambiguous diagnostic results cannot be enrolled in the study. If the ADOS-2 assessment has been performed by a certified rater and documented within 12 months of the screening visit, it is not mandatory to repeat it unless the subject was assessed below an age of 2 years.
* Hearing and vision compatible with the study assessments, as judged by the investigator
* Ability for subject and the caregiver to comply with the study protocol, in the investigator's judgment
* Availability of a parent or other reliable caregiver who is fluent in language of the site and has frequent and sufficient contact with the subject.

Exclusion Criteria:

* Clinically significant psychiatric and/or neurologic comorbidity that may interfere with the safety or efficacy endpoints in the view of the investigator
* Clinically significant regression of any acquired language and motor function skills in the opinion of the investigator throughout the subject's development
* History of seizures with the exception of a single, non-complicated febrile seizure >= 6 months before screening
* Clinical diagnosis of peripheral neuropathy or signs and symptoms indicative of peripheral neuropathy
* Any clinically relevant cardiovascular disease
* Confirmed elevation in cardiac troponin I (cTn I), high-sensitive cardiac troponin T (hs cTn T), N-terminal pro-B-type natriuretic peptide (NT-proBNP) or, if conducted, clinically relevant abnormality in Doppler echocardiogram
* Confirmed clinically significant abnormality on ECG at screening, including, but not limited to, a QT interval corrected through use of Fridericia's formula (QTcF) of >= 450 ms, absence of dominating sinus rhythm, or second- or third-degree atrioventricular block
* Confirmed systolic or diastolic blood pressure above the 95th percentile or below the 5th percentile according to the Centers for Disease Control and Prevention (CDC) norm tables referring to stature (height)-for-age percentiles
* Confirmed heart rate: >150 bpm in 2-year old children, >135 bpm in 3-year old children, or >120 bpm in 4-year old children.
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study; or discontinuation of prohibited medication that might pose unacceptable risks to the subject in the opinion of the investigator
* Evidence for current GI disease that would interfere with the conduct of the study or pose unacceptable risks in the opinion of the investigator
* History of coagulopathies, bleeding disorders, or blood dyscrasias
* Positive serology for HIV-1 or HIV-2
* Confirmed clinically significant abnormality in parameters of hematology, clinical chemistry, coagulation, or urinalysis, specifically a confirmed absolute neutrophil count (ANC) <LLN Children with confirmed CPK elevations exceeding 2 x upper limit of normal (ULN) will be excluded
* History of malignancy
* Clinically significant loss of blood within 3 months prior to screening
* Unstable use of permitted medications for 4 weeks before screening
* Use of prohibited medications within 30 days (or 5 times the half-life, whichever is longer) prior to initiation of study treatment

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (5):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - Richmond Behavioral Associates, Staten Island, New York
  - University Hospitals Cleveland Medical Center; Division of Child and Adolescent Psychiatry, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Red Oak Psychiatry Associates, PA, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Balovaptan
Started | 2
Completed | 1
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Balovaptan
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.45 (0.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve at Steady State (AUCss) of Balovaptan
Time Frame: Predose, 2, 4, 6 hours postdose at Week 2; predose at Week 6; predose at Week 12; predose at Week 24, predose at Week 54
Population: Due to low enrollment number patient analysis are not provided to protect participant confidentiality.
Arm/Group | Balovaptan
Number analyzed (Participants) | 0

2. Primary Outcome: Plasma Concentration of Balovaptan
Time Frame: as for outcome 1
Population: Due to low enrollment number patient analysis are not provided to protect participant confidentiality.
Arm/Group | Balovaptan
Number analyzed (Participants) | 0

3. Primary Outcome: Plasma Concentration of M2 Metabolite, as Applicable
Time Frame: as for outcome 1
Population: Due to low enrollment number patient analysis are not provided to protect participant confidentiality.
Arm/Group | Balovaptan
Number analyzed (Participants) | 0

4. Primary Outcome: Plasma Concentation of M3 Metabolite
Time Frame: as for outcome 1
Population: Due to low enrollment number patient analysis are not provided to protect participant confidentiality.
Arm/Group | Balovaptan
Number analyzed (Participants) | 0

5. Primary Outcome: Plasma Concentration Ratio of M2 to Balovaptan, as Applicable
Time Frame: as for outcome 1
Population: Due to low enrollment number patient analysis are not provided to protect participant confidentiality.
Arm/Group | Balovaptan
Number analyzed (Participants) | 0

6. Primary Outcome: Plasma Concentration Ratio of M3 to Balovaptan
Time Frame: as for outcome 1
Population: Due to low enrollment number patient analysis are not provided to protect participant confidentiality.
Arm/Group | Balovaptan
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Up to approximately week 20
Measure: Number; unit: Number of Participants
Arm/Group | Balovaptan
Number analyzed (Participants) | 2
Number of Participants | 2

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 6 May 2020 (up to approximately 20 weeks)
Description: The safety population is defined as patients who received any amount of study treatment.
Arm/Group | Balovaptan
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balovaptan (N=2)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated with 2 participants enrolled. Due to low enrollment number patient analysis are not provided to protect participant confidentiality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT04049578/Prot_SAP_000.pdf